CLINICAL TRIAL: NCT02300324
Title: An Intervention Study to Assess the Bioavailability of Sulforaphane Delivered by Glucoraphanin-enriched Broccoli Soups in Healthy Subjects
Brief Title: The Bioavailability Of Sulforaphane From Broccoli Soups Study (BOBS)
Acronym: BOBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: Biotechnology and Biological Sciences Research Council (Other); Prostate Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 14/EE/1121
Record Dates: First submitted 2014-11-20; First posted 2014-11-25 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Healthy
Keywords: bioavailability; Beneforte; sulforaphane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Standard v Beneforte v Beneforte Extra (Experimental): This is a randomized, double-blinded, three-phase crossover trial investigating the bioavailability of SF following consumption of three types of broccoli + stilton soup containing different concentrations of glucoraphanin. The three types of soup are standard broccoli and stilton soup, beneforte broccoli and stilton soup, and beneforte extra broccoli and stilton soup.
  Interventions: Dietary Supplement: Standard broccoli and stilton soup; Dietary Supplement: Beneforte broccoli and stilton soup; Dietary Supplement: Beneforte Extra broccoli and stilton soup

INTERVENTIONS:
Dietary Supplement: Standard broccoli and stilton soup — Participants will be randomised to eat one portion (300g) of broccoli soup for each phase.
Dietary Supplement: Beneforte broccoli and stilton soup — Participants will be randomised to eat one portion (300g) of broccoli soup for each phase.
Dietary Supplement: Beneforte Extra broccoli and stilton soup — Participants will be randomised to eat one portion (300g) of broccoli soup for each phase.

SUMMARY:
There is current evidence that suggests eating cruciferous vegetables like broccoli, cauliflower, cabbage is beneficial to our health as they contain compounds which are thought to reduce the risk of diseases such as cancer and cardiovascular diseases. Cruciferous vegetables are able to deliver in our body a group of compounds called isothiocyanates (ITCs) that are thought to be responsible of their health-promoting effects. Sulforaphane (SF) from broccoli is one of the most studied ITCs and its anticancer properties have been extensively investigated in in vitro and in vivo models.

The investigators propose to undertake an intervention study to measure the bioavailability of SF from the soups used in another intervention study called ESCAPE. The investigators would like to investigate the rate and extent to which SF reaches the systemic circulation and is excreted in urine by measuring SF and its metabolites in plasma and urine samples collected from apparently healthy participants after consumption of the three types of broccoli + stilton soups. The three types of soups are standard broccoli + stilton soups and two high-glucoraphanin (SF precursor) broccoli + stilton soups which are able to deliver different levels of SF.

This study has been funded by Biotechnology and Biological Sciences Research Council (BBSRC) and Prostate Cancer foundation (PCF).

DETAILED DESCRIPTION:
This study will be a randomized, double-blinded, three-phase crossover trial which will investigate the bioavailability of SF following consumption of broccoli + stilton soup containing different concentrations of glucoraphanin.

The study population will consist of non-smoking men and women aged between 18 and 65 years old. Participants will undergo three phases separated by a minimum of two weeks (wash-out period). Each phase will consist of a 48 hour pre-intervention diet restriction, a study day involving an 8 hour cannulation at the Human Nutrition Unit (HNU) of the Institute of Food Research (IFR) and collection of a 24 hour urine and blood sample the following morning. Participants will be randomly allocated to one of the three soups in each phase. The following soups will be tested in the three phases: i) 300g standard broccoli + stilton soup, ii) 300g Beneforte® broccoli + stilton soup, iii) 300g Beneforte Extra broccoli + stilton soup.

Beneforte and Beneforte extra broccoli are especially cultivated to deliver high sulforaphane levels after consumption. All the three broccoli varieties have the same appearance and flavour thus enabling a blinded human intervention study to be undertaken. Broccoli soups will be manufactured by a food company that supplies soups to the leading supermarket retailers in the United Kingdom.

Each phase will consist of a 48 hour pre-intervention diet restriction, a study day (study day 1) comprising of approximately a nine hour stay at the HNU which will involve cannulation. The following morning participants will visit the HNU for up to 1 hour for collection of a single blood sample at 24 hour post-dose followed by breakfast. During study day 1, eleven 10ml blood samples will be collected over the course of the day from participants at the following timepoints: 0, 30, 45, 60, 90, 120, 180, 240, 360, 480 mins and a 24 hour blood sample. Six urine samples will be collected at the following timepoints: 0, 0-2, 2-4, 4-6, 6-8, 8-24 hours.

The three phases will be separated by a minimum of a two week washout period. For the duration of the study, participants will be required to follow a glucosinolate-free diet for a total of nine days which will be three days per phase. The three days are split into 48 hours (2 days) prior to the study day, 24 hours (1 day) on the study day as well as the following morning until the 24 hour blood and urine sample have been collected. After the 24 hour urine and blood samples have been collected, participants can resume their normal diet for a minimum of two weeks until 48 hours prior to their next study day. This will reduce the contribution of glucosinolate from other foods having an impact on the results of the study. The involvement of the participants will last approximately 11-12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Aged 18-65 years
* Non-smokers
* Those that live within 40 miles of IFR
* Those who like broccoli + stilton soups

Exclusion Criteria:

* Those unwilling/unable to provide urine and blood samples
* Results of the clinical screening indicate, or are judged by the HNU medical advisor to be indicative of a health problem which could compromise the well-being of the participants if they participated, or which would affect the study outcome.
* Those whose vein status is assessed by HNU senior research nurse as unsuitable for cannulation
* Known history of fainting when blood samples are taken, feel unwell or faint during any clinical study day procedures at the HNU
* Women who are or have been pregnant within the last 12 months or who are breast feeding.
* Those diagnosed with any long-term medical condition (e.g. diabetes, haemophilia, cardiovascular disease, glaucoma, anaemia) or requiring medication that may affect the study outcome.
* Smokers
* Those taking dietary supplements or herbal remedies which may affect the study outcome - unless the participant is willing to discontinue taking them for 1 month prior to starting study. Please note that some supplements may not affect the study and this will be assessed on an individual basis
* Those allergic to any of the ingredients in broccoli + stilton soups
* Participants allergic to members of the Brassica family, e.g. mustard allergy (often combined with sensitivity to mugwort pollen, cabbage and peach) or to Brassica pollens (mustard or rapeseed).
* Those taking any prescribed or non-prescribed medication (short or long term), which may affect the study data or participant's wellbeing. This will be assessed by the HNU medical advisor on an individual basis.
* Those on an anti-coagulant therapy or have had anti-coagulant therapy in the past 3 months.
* Parallel participation in another research project that involves dietary intervention
* Any person related to or living with any member of the study team
* Participation in another research project, which involves blood sampling within the last four months unless total blood from both studies does not exceed 470mL (unless the participants are willing to wait 4 months and then be re-screened).
* Those unwilling to provide GP's contact details
* Those unable to provide written informed consent
* Those not suitable to take part in this study because of the screening results
* Those who have donated or intend to donate blood within 16 weeks prior to the study or during the study
* Those with a body mass index (BMI, kg/m2) ≤20 or ≥35 kg/m2
* Depressed or elevated blood pressure measurements (<90/50 or 95/55 if symptomatic or >160/100)
* Those that have used antibiotics within the previous one month or on long-term antibiotic therapy.
* Those who are unable to completely finish the 300g portion of broccoli + stilton soup on any of the study days as this will affect study data.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Total excretion of SF in 24 hour urine samples | 0, 0-2, 2-4, 4-6, 6-8, 8-24 hours
  To measure the total excretion of SF in urine collected for 24 hours after consumption of one pot (300g) of three types of broccoli + stilton soup containing different concentrations of glucoraphanin, SF precursor.

SECONDARY OUTCOMES:
Plasma concentration of SF and its metabolites | 0, 30, 45, 60, 90, 120, 180, 240, 360, 480 mins and 24 hours
  • To measure SF and its metabolites in plasma following consumption of one pot (300g) of three types of broccoli + stilton soup containing different concentrations of glucoraphanin.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Mithen, PhD, Principal Investigator — Quadram Institute Bioscience
Locations (1):
- Institute of Food Research, Norwich, Norfolk, United Kingdom

REFERENCES:
- [Derived] Sivapalan T, Melchini A, Saha S, Needs PW, Traka MH, Tapp H, Dainty JR, Mithen RF. Bioavailability of Glucoraphanin and Sulforaphane from High-Glucoraphanin Broccoli. Mol Nutr Food Res. 2018 Sep;62(18):e1700911. doi: 10.1002/mnfr.201700911. Epub 2018 Mar 8. PMID 29266773